CLINICAL TRIAL: NCT02978456
Title: Quantitative Coronary Angiography Versus Intravascular Ultrasound GUIDancE for Drug-Eluting Stent Implantation: GUIDE-DES Trial
Brief Title: Quantitative Coronary Angiography Versus Intravascular Ultrasound GUIDancE for Drug-Eluting Stent Implantation
Acronym: GUIDE DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, professor, Division of Cardiology, Department of Internal Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-24
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Coronary Disease; Coronary Stenoses
Keywords: IVUS guided PCI; QCA guided PCI
MeSH Terms: conditions — Coronary Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quantitative coronary angiography guided (Experimental)
  Interventions: Device: quantitative coronary angiography guided coronary intervention with sirolimus-eluting Orsiro/Orsiro mission stent
- Intravascular ultrasound guided (Active Comparator)
  Interventions: Device: intravascular ultrasound guided coronary intervention with sirolimus-eluting Orsiro/Orsiro mission stent

INTERVENTIONS:
Device: quantitative coronary angiography guided coronary intervention with sirolimus-eluting Orsiro/Orsiro mission stent — In the quantitative coronary angiography-guided group, sirolimus-eluting Orsiro/Orsiro mission stent size and length is chosen to cover the entire length of the culprit lesions according to quantitative coronary angiography measurements. Selection of the sirolimus-eluting Orsiro/Orsiro mission stent size should be guided by both quantitative coronary angiography measurement and visual estimate, and is recommended to be based on distal reference vessel diameter by quantitative coronary angiography (distal reference vessel diameter by quantitative coronary angiography plus ~10% of distal reference vessel diameter).
  Arms: quantitative coronary angiography guided
Device: intravascular ultrasound guided coronary intervention with sirolimus-eluting Orsiro/Orsiro mission stent — In the intravascular ultrasound -guided group, sirolimus-eluting Orsiro/Orsiro mission stent size and length is selected by intravascular ultrasound measurements.
  Arms: Intravascular ultrasound guided

SUMMARY:
The purpose of this study is to compare clinical outcomes between quantitative coronary angiography -guided and Intravascular ultrasound -guided strategy in patients with significant coronary artery disease undergoing sirolimus-eluting Orsiro/Orsiro mission stent implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 19years of age
2. Typical chest pain or objective evidence of myocardial ischemia suitable for elective PCI
3. Significant coronary artery lesions suitable for sirolimus-eluting Orsiro/Orsiro mission stent implantation
4. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Angiographic exclusion criteria: any of the followings 1)Bypass graft lesions 2)Impaired delivery of IVUS is expected:

   * Extreme angulation (≥90°) proximal to or within the target lesion.
   * Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   * Heavy calcification proximal to or within the target lesion.
2. Previous percutaneous coronary intervention within 6 months before the index procedure
3. Previous BVS (bioresorbable vascular scaffold) implantation
4. Left ventricular ejection fraction (LVEF) < 30%
5. Hypersensitivity or contraindication to device material and its degradants and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated.
6. Persistent thrombocytopenia (platelet count <100,000/µl)
7. Any history of hemorrhagic stroke or intracranial hemorrhage, Transient ischemic attack or ischemic stroke within the past 6 months
8. A known intolerance to antiplatelet agents (aspirin, clopidogrel, prasugrel or ticagrelor)
9. Any surgery requiring general anesthesia or discontinuation of aspirin and/or an ADP antagonist is planned within 12 months after the procedure.
10. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
11. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
12. Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
13. Life expectancy < 1 years for any non-cardiac or cardiac causes
14. Unwillingness or inability to comply with the procedures described in this protocol.
15. Patient's pregnant or breast-feeding or child-bearing potential.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1528 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 12 months
  the cumulative incidence of cardiac death, target vessel myocardial infarction or ischemia-driven target lesion revascularization at 12 months after the index procedure.

SECONDARY OUTCOMES:
Procedural success | 24 hours
  Achievement of final stent residual stenosis of less than 30% by QCA with successful deployment of at least one stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (24 hour after an index procedure).
Death (cardiac, vascular, non-cardiovascular) | 12 months
Myocardial infarction | 12 months
Stent thrombosis (definite/probable) | 12 months
Stroke | 12 months
Target lesion revascularization | 12 months
Any revascularization | 12 months
Economic analysis | 12 months
  cost-effectiveness of QCA- versus IVUS-guided DES implantation

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Korea University Anam Hospital, Anam
  - Hallym University Medical Center, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Asan Medical Center, Seoul
  - Gangnam Severance Christian Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee PH, Hong SJ, Kim HS, Yoon YW, Lee JY, Oh SJ, Lee JS, Kang SJ, Kim YH, Park SW, Lee SW, Lee CW; GUIDE-DES Trial Research Group. Quantitative Coronary Angiography vs Intravascular Ultrasonography to Guide Drug-Eluting Stent Implantation: A Randomized Clinical Trial. JAMA Cardiol. 2024 May 1;9(5):428-435. doi: 10.1001/jamacardio.2024.0059. PMID 38477913
- [Derived] Lee PH, Hong SJ, Kim HS, Yoon YW, Lee JY, Oh SJ, Kang SJ, Kim YH, Park SW, Lee SW, Lee CW; GUIDE-DES Trial Research Group. Quantitative coronary angiography versus intravascular ultrasound guidance for drug-eluting stent implantation (GUIDE-DES): study protocol for a randomised controlled non-inferiority trial. BMJ Open. 2022 Jan 13;12(1):e052215. doi: 10.1136/bmjopen-2021-052215. PMID 35027418